CLINICAL TRIAL: NCT04254055
Title: Effectiveness of a Training Program Through Plyometric, Proprioceptive and Strength Exercises in Order to Observe an Improvement of the Strength, Stability and Functional Stability of the Shoulder in Rugby Players
Brief Title: Plyometric, Proprioceptive and Strength Exercises in Rugby Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEF
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Overhead Athletes
Keywords: Shoulder; Strength; Stability; Functionality; Rugby.
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Exercise 1 with medicine ball. Standing player with 90º shoulder abduction and elbow flexion. He will receive the ball with an external rotation returning it with internal rotation. Exercise 2 with elastic band. From standing, he will fix the elastic band with his foot and perform a shoulder flexion with his contralateral limb. Exercise 3 of iron with support of the hands on the floor and shoulder, elbow and wrist aligned. You should perform a scapula approach and separation without altering its initial position. Exercise 4 BodyBlade ©. From standing with 90º of 90 ° shoulder abduction and elbow flexion. It will perform an anteroposterior thrust, causing a wave effect to stabilize the shoulder joint for 30 seconds.
  Athletes will do 15 repetitions of each exercise.
  Interventions: Other: exercises
- Control group (No Intervention): Players included in the control group will not receive any intervention.

INTERVENTIONS:
Other: exercises — Those subjects included in the experimental group will receive an intervention through a program with plyometric, proprioceptive and strength exercises. The subjects included in the control group will not receive any intervention.
  Other Names: Experimental group
  Arms: Experimental group

SUMMARY:
Introduction. Shoulder injury is the pathology that causes the longest downtime in rugby players, representing 66% of upper limb injuries in this discipline. The lack of strength, and instability are factors that predispose the athlete to suffer this type of dysfunction. The intervention of the study consists of a training program that counteract these dysfunctions.

Aim. Assess the effectiveness of a program using plyometric, proprioceptive and strength exercises on 18-45-year-old rugby players to improve strength and stability.

Study design. Clinical randomized, prospective, single-blind and trackable. Methods. The subjects included in two study groups, experimental and control, will be attributed a random order. The treatment will last 4 weeks, with 2 weekly sessions, of approximately 25 minutes each. The study variables will be strength, stability and functionality. A descriptive statistical analysis will be carried out calculating the main statistical characteristics. Through of a Kolmogorov analysis the normality of the sample will be assessed. A t-Student test for paired samples will be performed for the difference between the means of the dependent and independent variables. An analysis if variance (ANOVA) for repeated measures will be used to compare the means and checked to what extent the intra-subjects factors influence the dependent variables.

Expected results. Improved shoulder strength, stability and functionality for the subjects on which the study is carried out.

ELIGIBILITY:
Inclusion Criteria:

* Federated rugby players
* Male
* 18 to 45 years old
* Currently participating in regional competitions

Exclusion Criteria:

* Being treated with anti-inflammatory drugs
* Having suffered an upper limb injury in the month prior to the intervention
* Have undergone surgery for any shoulder pathology during the previous 12 months
* Who have suffered or suffer from a serious and / or metabolic disease
* That they have not signed the informed consent

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline strength after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The strength assessment will be carried out with a dynamometer. The subject will stand up and the examiner will indicate when the movement should begin. The dynamometer will be positioned to measure the strength of the shoulder abductors and rotators in the position of 90º of abduction and 90º of external rotation. The unit of measure is the Newton

SECONDARY OUTCOMES:
Change from baseline stability after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be assessed with the Closed Kinetic Chain Upper Extremity Stability Test. The initial position of the test is a push-up position with the upper extremities perpendicular to the ground. We will use two strips of 3.80 cm tape stuck on the floor and separated 91.44cm apart. The subjects will carry one of the hands until they touch the other strip of tape and return to the initial position. The touches will be counted every time one of the tape strips is touched in a total time of 15 seconds. Each subject will perform a warm-up, followed by 3 attempts with a break between attempts, of 45 seconds, averaging the 3 data obtained.
Change from baseline functionality after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment will be carried out with the Simple Shoulder Test. This test is a questionnaire of 12 questions, with two answer options: yes (when the subject is able to perform the task) and no (when he is not able to do it). The results obtained have a scoring range from 0 to 12, with 0 being the lowest functionality and 12 being the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- European University of Madrid, Madrid, Spain